CLINICAL TRIAL: NCT00601289
Title: An Open Label, Multicenter, Phase II Study Evaluating the Safety and Efficacy of Temozolomide Treatment in Patients With Invasive Pituitary Tumors
Brief Title: Temozolomide in Treating Patients With Invasive Pituitary Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding term ended
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000577534; 07-05-077-01
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: pituitary chromophobe adenoma; recurrent pituitary tumor; ACTH-producing pituitary tumor; growth hormone-producing pituitary tumor; prolactin-producing pituitary tumor; pituitary basophilic adenoma; pituitary eosinophilic adenoma; prolactin secreting adenoma; nonfunctioning pituitary tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Adenoma, Chromophobe; Pituitary Neoplasms; Growth Hormone-Secreting Pituitary Adenoma; Adenoma, Basophil; Adenoma, Acidophil; Prolactinoma | interventions — Temozolomide; DNA Methylation; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: temozolomide
Genetic: DNA methylation analysis
Genetic: microarray analysis
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with invasive pituitary tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of temozolomide on pituitary tumor growth in patients with invasive pituitary tumors.
* To assess the effect of temozolomide on pituitary tumor response and the duration of tumor response in these patients.

Secondary

* To assess the effect of temozolomide on pituitary tumor hormone secretion in these patients.
* To assess the effect of temozolomide on other aspects of pituitary function in these patients.
* To assess the overall safety and tolerability of temozolomide in these patients.
* To assess the overall quality of life of patients treated with temozolomide.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of 12 courses, patients achieving a complete or partial tumor response may continue to receive temozolomide at the investigator's discretion in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected periodically to assess methylation status of the methyl-guanine methyl-transferase promoter (MGMT) gene and to quantitate immunocytochemical expression of the tumor suppressor proteins p53, p16, and p27. Tissue samples are also analyzed by microarray and proteomics to determine a genetic "signature" of invasive vs non-invasive pituitary tumors and to determine if this signature correlates with response to temozolomide. Blood samples are also periodically for biomarker laboratory studies.

Patients complete a quality of life questionnaire periodically.

After completion of study therapy, patients are followed for 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically demonstrable invasive pituitary macroadenoma, including any of the following subtypes:

  * Growth hormone-secreting
  * Prolactin-secreting
  * Adrenocorticotrophic hormone-secreting
  * Non-secreting
* Must have biochemical evidence of any of the following:

  * Acromegaly as measured by serum insulin-like growth factor-1 (IGF-1)
  * Prolactinoma as measured by serum prolactin (PRL)
  * Cushing's disease as measured by 24-hour urinary-free cortisol
* Inadequate tumor control, defined as a visible pituitary tumor ≥ 1 cm in maximal diameter encasing the carotid arteries, and/or invading into the cavernous sinuses, and/or abutting/invading the optic chiasma as demonstrated by MRI scan with or without contrast
* Previously assessed by radiosurgery and meets ≥ 1 of the following criteria:

  * Not a suitable candidate for radiotherapy (e.g., tumor abutting and/or invading the optic chiasm)
  * Declined radiotherapy (in light of side effects or personal choice)
  * Has not exhibited tumor shrinkage or tumor continues to grow ≥ 1 year after completion of radiotherapy
* Must have a normal visual field evaluation by Goldman perimetry

  * No visual field abnormalities
* Hypopituitarism allowed as evidenced by any or all of the following:

  * Subnormal growth hormone response to arginine/growth hormone-releasing hormone testing (normal response is an increase of > 4 ng/mL)
  * Low age- and sex-matched IGF-1 levels
  * Low thyroid-stimulating hormone (TSH), free triiodothyronine (T3), and free thyroxine (T4) levels
  * Low estradiol levels
  * Low luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in postmenopausal female patients OR low testosterone, LH, and FSH levels in male patients
  * Serum cortisol < 3 ng/mL (at 8 am)
* Patients diagnosed with hypopituitarism (except for post-menopausal females) are required to initiate hormone replacement therapy for the 12-month duration of the study and to discontinue hormone replacement therapy at the end of 12 months to re-evaluate hypopituitarism

PATIENT CHARACTERISTICS:

* Able to undergo a pituitary MRI scan
* No clinically significant renal, hematologic, or hepatic abnormalities
* No prior or concurrent medical condition that may interfere with the conduct of the study or the evaluation of its results, in the opinion of the Investigator or the Data Safety Monitoring Board compliance officer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 2 months prior to, during, and for 1 month after completion of study therapy
* No history of immunocompromise, including known HIV positivity as measured by enzyme linked immunosorbent assay (ELISA) and western blot
* No alcohol or drug abuse within the past 6 months
* No blood donation within the past 2 months
* No history of noncompliance to medical regimens, potential unreliability, or inability to complete the entire study
* No other active malignant disease within the past 5 years, except basal cell carcinoma or carcinoma in situ of the cervix
* No active or suspected acute or chronic uncontrolled infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior pituitary surgery allowed provided the surgery failed to induce complete tumor response and the patient is deemed unsuitable for further pituitary surgeries
* At least 3 months since prior pituitary surgery
* More than 1 month since prior unlicensed drugs or participation in a clinical trial with an investigational drug
* No concurrent pituitary surgery or pituitary radiotherapy
* No other concurrent therapy to reduce pituitary tumor size

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pituitary tumor control as assessed by MRI at 3, 6, 9, and 12 months | 1 year
Change in Tumor response rate (complete response or partial response) from baseline as assessed by RECIST criteria at 3, 6, 9, and 12 months | 1 year
Rebound tumor growth as assessed by MRI at 6 months after completion of treatment | 6 months

SECONDARY OUTCOMES:
Biochemical control as assessed by measurement of hormones secreted in excess by the pituitary tumor at baseline, at 3, 6, 9, and 12 months during treatment, and then at 2 months after completion of treatment | 14 months
Pituitary function as assessed by standard pituitary function tests at baseline and at 6 months and 12 months | 1 year
Safety and tolerability of temozolomide as assessed by NCI CTC v2.0 at screening, baseline, and then monthly until study completion | 1 year
Overall quality of life as assessed by Karnofsky performance status questionnaire periodically during study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Heaney, MD, Study Chair — Jonsson Comprehensive Cancer Center